CLINICAL TRIAL: NCT02133404
Title: Phase II Study of ASP7991 -A Double-blind, Cinacalcet Hydrochloride-controlled, Dose-ascending Study in Secondary Hyperparathyroidism Patients Undergoing Hemodialysis -
Brief Title: A Study to Evaluate the Effect of ASP7991 in Secondary Hyperparathyroidism Patients Undergoing Hemodialysis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7991-CL-1004
Record Dates: First submitted 2014-04-29; First posted 2014-05-08 (Estimated); Last update posted 2024-11-06 (Actual); Status verified 2024-10

CONDITIONS: Secondary Hyperparathyroidism
Keywords: Mineral bone disease(MBD); Chronic kidney disease(CKD); secondary hyperparathyroidism(SHPT)
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Renal Insufficiency, Chronic | interventions — ASP7991; Cinacalcet

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ASP7991 group (Experimental): receiving ASP7991 and Cinacalcet-placebo
  Interventions: Drug: ASP7991; Drug: Placebo
- Cinacalcet group (Active Comparator): receiving Cinacalcet and ASP7991-placebo
  Interventions: Drug: Cinacalcet; Drug: Placebo

INTERVENTIONS:
Drug: ASP7991 — oral
  Arms: ASP7991 group
Drug: Cinacalcet — oral
  Arms: Cinacalcet group
Drug: Placebo — oral

SUMMARY:
To examine efficacy and safety after 12-week administration of ASP7991 in secondary hyperparathyroidism patients undergoing hemodialysis

DETAILED DESCRIPTION:
This study is a multicenter, double-blind, randomized, Cinacalcet hydrochloride-controlled, parallel-group, dose-ascending study. Subjects judged to be eligible will be registered and randomized into either ASP7991 group (receiving ASP7991 and cinacalcet-placebo) or Cinacalcet group (receiving cinacalcet and ASP7991-placebo), and will receive 12-week (84 days) administration of study drug from first dialysis day in a week (treatment period), in a double-blind manner. The dose of the study drugs will be increased every 3 weeks in dose-ascending manner.

Follow-up assessment will be performed before starting first dialysis in a week, 1 week (7 days) after the completion of the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are on stable chronic maintenance dialysis who are receiving hemodialysis therapy 3 times/week since before 12-week (84 days) administration and are also scheduled to undergo the regimen of 3 times/week hemodialysis during the study period
* Patients with secondary hyperparathyroidism
* Patients whose serum iPTH concentration is >240 pg/mL and corrected serum Ca is ≥ 9.0 mg/dL
* Patients who have had no changes in the following items ≥4-week (28 days).

  * Dosage and regimen, including new administration, of active vitamin D, calcitonin preparation, phosphate binder, and medication with phosphate absorption (including foods)
  * Ca concentration of the dialysate, membrane area of the dialyzer, and dialysis time of each week

Exclusion Criteria:

* Patients who underwent parathyroid intervention, such as parathyroidectomy (PTx) or percutaneous ethanol injection therapy (PEIT), within 24 weeks (168 days) prior to the administration
* Patients who have primary hyperparathyroidism
* Patients who received bisphosphonate, estrogen preparation, parathyroid hormone within 4 weeks (28 days)
* Patients with uncontrolled hypertension (systolic blood pressure ≥ 180 mmHg and diastolic blood pressure ≥ 120 mmHg are observed at >2/3 of all confirmable measurements
* Patients who are complicated by severe heart disorder [congestive cardiac failure (NYHA classification III or higher), or wide range of old myocardial infarction], or having a history of hospitalization for cerebro-vascular disease or heart disorder within 12 weeks (84 days) before administration of the study drug
* Patients with hepatic function abnormal (ALT or AST is >2× ULN, or total bilirubin (T-bil) is > 1.5 × ULN.)
* Patients with a history of malignant tumor or the patient's condition is complicated by malignant tumor. (However, enrollment is acceptable if the tumor has not relapsed for 5 years or longer.)
* Patients with a history of serious drug allergy including anaphylactic shock
* Patients with a history of drug allergy to Cinacalcet hydrochloride
* Female patients who are potentially child-bearing or lactating, or patients who do not comply with the instructed contraceptive measures
* Patients who were or are currently involved in trials for other investigational drugs or medical devices, or clinical trial for post-marketing study drugs within 12 weeks (84 days) before the study
* Patients who have received ASP7991 in the past
* Patients who were judged ineligible to participate in the study by the

investigator / subinvestigator

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2014-03-14 (Actual); Primary Completion 2014-11-10 (Actual); Study Completion 2014-11-10 (Actual)

PRIMARY OUTCOMES:
Serum iPTH concentration | Before and at 8, 15, 22, 24, 29, 36, 43, 45, 50, 57, 64, 66, 71, 78, 85 and 92 days after start of the treatment
  iPTH: intact parathyroid hormone

SECONDARY OUTCOMES:
Corrected serum Ca, Phosphate(P) concentration | Before and at 3, 8, 15, 22, 24, 29, 36, 43, 45, 50, 57, 64, 66, 71, 78, 85 and 92 days after start of the treatment
  Ca x P will be calculated
serum vitamin D concentration | Before and at 22, 43, 64, 85 and 92 days after start of the treatment
serum wPTH concentration | Before and at 22, 43, 64, 85 and 92 days after start of the treatment
  wPTH: whole parathyroid hormone
Serum concentration of bone metabolism markers | Before and at 22, 43, 64, 85 and 92 days after start of the treatment
  Bone metabolism markers will be BAP (Bone specific alkaline phosphatase) and TRACP5b (Tartrate-resistant acid phosphatase-5b)
Serum FGF23 concentration | Before and at 22, 43, 64, 85 and 92 days after start of the treatment
Safety assessed by the incidence of adverse events, vital signs, laboratory tests and 12-lead ECGs | For 12 weeks after start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (6):
- Japan (6):
  - Chugoku
  - Chūbu
  - Kanto
  - Kyushu
  - Shikoku
  - Tōhoku

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results Web site — https://astellasclinicalstudyresults.com/study.aspx?ID=277